CLINICAL TRIAL: NCT02390583
Title: Internet Addiction and Sleep Disorders
Acronym: ADDICSOM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120140
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Internet Addiction
Keywords: Internet dependence; Sleep disorders; pathological gambling
MeSH Terms: conditions — Internet Addiction Disorder; Sleep Wake Disorders; Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): CBT treatment of internet dependence each two weeks during 3 months
  Interventions: Behavioral: CBT treatment of internet dependence
- intervention (Experimental): CBT treatment of internet dependence plus CBT treatment of sleep disorders during 3 months
  Interventions: Behavioral: CBT treatment of internet dependence; Behavioral: CBT treatment of sleep disorders

INTERVENTIONS:
Behavioral: CBT treatment of internet dependence — CBT treatment of internet dependence
Behavioral: CBT treatment of sleep disorders — CBT treatment of sleep disorders
  Arms: intervention

SUMMARY:
This is an open label randomized controlled trial, comparing two modes of treatment for internet addiction (gaming or gambling online) with sleep disorders associated.

DETAILED DESCRIPTION:
We will check sleep disorders among patients presenting internet dependence. Diagnosis will be followed by a specific treatment during three months. This treatment is expected to reduce prevalence of internet dependence and associated addictive disorders (alchohol, nicotine) . rate of sleep disorders is also expected to decrease under treatment.

This is an open label randomized controlled trial, comparing two modes of treatment for internet addiction (gaming or gambling online) with sleep disorders associated.

Patients will be randomised in two arms : controls (CBT treatment of Internet dependence) and intervention (CBT treatment of addiction plus CBT treatment of sleep disorders).

ELIGIBILITY:
Inclusion Criteria:

* Internet addiction (Young scale ≥5)
* Online compulsive gambling ( DSM IV scale for pathological gambling and SOGS) and/or addiction to online gaming (problem video game playing ≥ 5)
* sleep latency >45 min/night and more than 3 nights a week
* subjective total sleep time <6h30/night more than 3 nights a week
* Adult patient

Exclusion Criteria:

* cognitive impairments, memory disorders, non french-speaking patients
* already known and on treatment sleep pathologies
* somatic conditions non compatible with clinical evaluation
* cybersex dependance
* Treatment with dopaminergic agents
* patients under jurisdictional assistance
* patients non covered by the french health system
* non consenting patients
* History of Healthcare for internet dependence
* Patients already treated for internet dependance
* pregnant or lactating women
* Patients already participating in other studies on internet dependance and sleeping disorders
* suicide attempt before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
number of hours each week spent gaming or online gambling | 6 months
  The evaluation period will be 7 days of follow-up visit at 6 months. Each patient will complete a connection agenda that will provide the therapist during follow-up visits.

SECONDARY OUTCOMES:
Number of hours spent on line gaming or online gambling | 3 months
insomnia | 3 and 6months
  measure with Insomnia Severity Index (ISI)
daytime sleepiness | 3 and 6 months
  daytime sleepiness with specific scales ( Epworth and KAROLINSKA)
total sleep time | 3 and 6 months
  total sleep time (actimetry, sleep agenda) Actimetry results will be centrally reviewed by experts blinded to realization date
number of awakenings during night | 3 and 6 months
  number of awakenings during night (actimetry) Actimetry results will be centrally reviewed by experts blinded to realization date
treatment with hypnotics | 3 and 6 months
  Number of tablets taken each week
Depression | 3 and 6 months
  score of depression at the MINI questionnaire
Anxiety | 3and 6 months
  Anxiety scores at the MINI questionnaire
Alcohol dependence | 3 and 6 months
  Alcohol dependence assess with severity AUDIT scale
Nicotine Dependence | 3 and 6 months
  assess with Fagerstrom scale
Other psychoactive agents | 3 and 6 months
  assess with RDAPS questionnaire
Compliance | 3 and 6 months
  Compliance will be studied with the participation of patients to CBT groups at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lejoyeux Lejoyeux, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat-Claude.Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No
At the end of the study, patient could be informed of result of the study if they wish.
  No individual result will be communicate.